CLINICAL TRIAL: NCT05948293
Title: Randomized Investigation With an AI Powered Medical Device to Select the First Dose of FSH for Controlled Ovarian Stimulation
Brief Title: FSH Doser for Controlled Ovarian Stimulation
Acronym: ALGO3
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Seeking financial support.
Sponsor: Clínica EUGIN (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALGO3
Record Dates: First submitted 2023-07-06; First posted 2023-07-17 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Infertility
Keywords: controlled ovarian stimulation; Follicle Stimulating Hormone; AI
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to arm allocation. The research team will also be blinded, with the exception of the data coordinator. The medical team, with the exception of the ones assigned to care for the participants, will also be blinded to arm allocation. The embryology laboratory team will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): In the intervention arm the first dose of FSH will be assigned by a machine learning model called IDoser.
  Interventions: Device: Machine learning model called IDoser
- Control arm (Active Comparator): In the control arm the first dose of FSH will be determined by the clinician following standard practice.
  Interventions: Procedure: Standard clinical practice

INTERVENTIONS:
Device: Machine learning model called IDoser — Patients in the intervention arm will be prescribed the first dose of FSH by IDoser, that will take into account the age of the patient, BMI, AFC and AMH. These data will be retrieved from the patient's clinical file after their first visit to the clinic, after providing the patient with informed consent documentation.
  Other Names: IDoserFSH
  Arms: Intervention arm
Procedure: Standard clinical practice — Patients in the control group will be prescribed their first dose of FSH by the clinician according to standard clinical practice.
  Arms: Control arm

SUMMARY:
The study aims to evaluate the effectiveness of an individualized FSH dosing model called IDoser in controlled ovarian stimulation (COS) for assisted reproduction. The randomized, controlled, multicenter trial involves 236 first cycle IVF patients, who will be assigned to either the intervention arm (using the IDoser model) or the control arm (standard clinician-determined dosing). The primary outcome is the number of mature oocytes retrieved, with the hypothesis of non-inferiority for the intervention arm. Secondary outcomes include cycle cancellations, risk of ovarian hyperstimulation syndrome (OHSS), and pregnancy and live birth rates.

ELIGIBILITY:
Inclusion Criteria:

* First IVF cycles
* Use of autologous oocytes
* Use of FSH on the first day of stimulation (which can be combined with luteinizing hormone, LH).

Exclusion Criteria:

* Natural ovarian stimulation cycles (without Controlled ovarian stimulation)
* Cycles where FSH is not measured in International Units (IU).

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of MII oocytes | 3 weeks (from enrollment to oocyte pick-up)
  Total number of mature MII oocytes retrieved at oocyte pick-up

SECONDARY OUTCOMES:
Cycle cancellation rate | 3 weeks (from enrollment to oocyte pick-up)
  Cycle cancellation rate defined as the number of patients with no MII oocytes at OPU divided by the total number of enrolled patients
OHSS risk | 3 weeks (from enrollment to oocyte pick-up)
  Risk of ovarian hyperstimulation defined as levels of estradiol > 5000 pg/ml and/or a number ≥ 18 follicles measuring ≥11mm at last ultrasound check
Clinical pregnancy rate | 10 weeks (from enrollment to detection of fetal heart beat)
  Clinical pregnancy rate defined as the detection of fetal heart beat observed at 7th week of gestation, per first embryo transfer
Live birth rate | 44 weeks (from enrollment to baby delivery)
  Live Birth rate, per first embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Mina Popovic, PhD, Principal Investigator — Eugin Group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Correa N, Cerquides J, Arcos JL, Vassena R, Popovic M. Personalizing the first dose of FSH for IVF/ICSI patients through machine learning: a non-inferiority study protocol for a multi-center randomized controlled trial. Trials. 2024 Jan 11;25(1):38. doi: 10.1186/s13063-024-07907-2. PMID 38212837